CLINICAL TRIAL: NCT00355082
Title: A Multicenter, Double-Blind, Randomized Conversion to Monotherapy Comparison of Two Doses of Lamotrigine for the Treatment of Partial Seizures
Brief Title: Conversion To Monotherapy With Lamictal Extended Release Tablets For Treatment Of Partial Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAM30055
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Epilepsy, Partial
Keywords: epilepsy; lamotrigine; Lamictal; monotherapy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lamotrigine 300 (Experimental): 300 mg/day treatment
  Interventions: Drug: lamotrigine, 300 mg/day
- lamotrigine 250 (Experimental): 250 mg/day treatment
  Interventions: Drug: lamotrigine, 250 mg/day

INTERVENTIONS:
Drug: lamotrigine, 300 mg/day — 300 mg/day
  Other Names: lamotrigine
  Arms: lamotrigine 300
Drug: lamotrigine, 250 mg/day — 250 mg/day
  Arms: lamotrigine 250

SUMMARY:
This study is being conducted to determine the effectiveness of a lower monotherapy dose of lamotrigine than that currently approved.

DETAILED DESCRIPTION:
The study consists of a Treatment phase, where efficacy is determined and a Continuation phase for extended safety information. The Continuation phase is open to all Treatment phase participants and those who did not qualify for treatment because of an insufficient number of seizures during the Baseline phase.

ELIGIBILITY:
Inclusion criteria:

* Male or Female ≥13 years of age
* Have a confident diagnosis of epilepsy with partial seizures for at least 24 weeks prior to the Baseline Phase
* Have a documented history of partial seizures such that the investigator must judge that the subject is likely to have at least 4 partial seizures during the 8-week Baseline Phase.
* Have experienced at least 4 partial seizures (i.e., simple or complex partial seizures with or without secondary generalization) during an 8-week (i.e., 56 days) prospective Baseline Phase with at least one partial seizure occurring during each 4-week (i.e., 28-day) period.
* NOTE: With prior authorization from GlaxoSmithKline (GSK), retrospective data may take the place of up to the first 4 weeks (i.e., first 28 days) of the Baseline Phase for subjects providing reliable documentation of the following:

  1. A complete daily seizure diary that includes the number, and type (i.e., simple or complex partial seizures with or without secondary generalization), of seizures experienced each day for up to 28 consecutive days immediately prior to the prospective Baseline Phase
  2. Stability of prescribed dosages of background antiepileptic drug (AED)
  3. Compliance with background AED

All subjects permitted to use retrospective baseline data must complete a minimum of four weeks (i.e., 28 days) of the prospective Baseline Phase. The retrospective plus the prospective Baseline Phases must equal the 56 consecutive days prior to the start of dosing with study drug.

* be currently receiving AED monotherapy treatment with a stable regimen of a non-enzyme inducing AED for at least four weeks prior to starting the Baseline Phase.
* be able and willing to maintain an accurate, complete, written daily seizure diary, or has a parent/caregiver who is able and willing to maintain and accurate, complete, written daily seizure diary for the entire duration of the study.
* be able to comply with the dosing of study drugs, background AED, and all study procedures.
* understand and sign written informed consent, or will have a parent or a legally authorized representative who has done so, prior to the performance of any study assessments
* if female, and of childbearing potential be using an acceptable form of birth control, to include one of the following:

  1. Complete abstinence from intercourse for two weeks before exposure to the study drug, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (a minimum of 2 weeks).
  2. Consistent and correct use of one of the following methods of birth control:

Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject.

Any intrauterine device (IUD) with a documented failure rate of less than 1% per year

Double barrier method consisting of spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm).

NOTE: Women who have had a hysterectomy, tubal ligation, or are post-menopausal are considered to be of non-childbearing potential.

NOTE: A pharmacokinetic interaction has been observed between lamotrigine (LTG) and estrogen-based oral contraceptives. Therefore, the use of hormonal therapy (e.g., for contraception or hormone replacement therapy) is not allowed.

Exclusion criteria:

* Exhibits any primary generalized seizures (e.g., absence, myoclonic primary generalized tonic-clonic seizures).
* Has had status epilepticus within the 24 weeks prior to, or during, the Baseline Phase.
* Is taking an enzyme-inducing AED (EIAED - e.g. carbamazepine, phenytoin, phenobarbital, primidone) or is taking more than 1 background AED.
* Is currently taking lamotrigine (LTG) or has previously had an adequate trial of LTG.
* Is currently taking felbamate
* Is using hormone therapy
* Is abusing alcohol and/or other substances
* Has taken an investigational drug within the previous 30 days or plans to take an investigational drug anytime during the study.
* Is receiving chronic treatment with any medication that could influence seizure control
* NOTE: Use of benzodiazepines is allowed as specified in Section 8.1.2
* Is currently following the ketogenic diet.
* Is using vagal nerve stimulation
* Is planning surgery to control seizures during the study.
* Is pregnant, breastfeeding, or planning to become pregnant during the study or within the three weeks after the last dose of study drug.
* Is suffering from acute or progressive neurological disease, severe psychiatric disease or severe mental abnormality that is likely to interfere with the objectives of the study.
* Has any clinically significant cardiac, renal, hepatic condition, or a condition that affects the absorption, distribution, metabolism or excretion of drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2006-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (59):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Loxahatchee Groves, Florida
  - GSK Investigational Site, Sunrise, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Flossmoor, Illinois
  - GSK Investigational Site, Urbana, Illinois
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, Pikesville, Maryland
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Cloud, Minnesota
  - GSK Investigational Site, Hattiesburg, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Vorhees, New Jersey
  - GSK Investigational Site, Lawrence, New York
  - GSK Investigational Site, Plainview, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Midvale, Utah
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Charleston, West Virginia
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (3):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Capital Fefderal, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Chile (2):
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, San José, Costa Rica
- GSK Investigational Site, San Juan, Puerto Rico, Puerto Rico
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Yekaterinburg
- South Korea (4):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Seoul
- Ukraine (10):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Luhansk
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Vinnitsa
  - GSK Investigational Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] French JA, Hammer AE, Vuong A, Messenheimer JA. Analysis of three lamotrigine extended-release clinical trials: comparison of pragmatic ITT and LOCF methodologies. Epilepsy Res. 2012 Aug;101(1-2):141-7. doi: 10.1016/j.eplepsyres.2012.03.015. Epub 2012 Apr 10. PMID 22497754
- [Background] French JA, Temkin NR, Shneker BF, Hammer AE, Caldwell PT, Messenheimer JA. Lamotrigine XR conversion to monotherapy: first study using a historical control group. Neurotherapeutics. 2012 Jan;9(1):176-84. doi: 10.1007/s13311-011-0088-3. PMID 22139591
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: LAM30055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LAM30055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LAM30055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LAM30055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM30055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LAM30055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LAM30055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants in the Treatment phase and all Baseline Failure participants are eligible to enter the Continuation phase. The Continuation phase is for long-term safety exposure to lamotrigine extended release (LTG XR) at 300 mg/day; it is not a cross-over phase.
Pre-assignment Details: The number of participants (par.) starting the Continuation phase (CP) does not equal the number completing the Treatment phase (TP), as 1) the CP was optional, 2) not everyone from the TP was eligible to enter the CP, and 3) par. who failed to qualify for the TP (Baseline Failures) were allowed to enter the CP. All par. start the TP at 300 mg/day.
Groups:
- Lamotrigine Extended-release (LTG XR), 300 mg: LTG XR, 300 mg/day. In the Continuation phase, Treatment phase participants received LTG XR, 300 mg/day.
- LTG XR, 250 mg: LTG XR, 250 mg/day
- Baseline Failures: Baseline failures that entered the Continuation Phase; LTG XR; 300 mg/day
Period: Double-Blind (DB) Treatment Phase
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg | LTG XR, 250 mg | Baseline Failures
Started | 113 (112 participants have baseline data; 1 participant did not receive study drug.) | 113 (111 participants have baseline data; 2 participants did not receive study drug.) | 0
Completed | 94 | 79 | 0
Not Completed | 19 | 34 | 0
Not completed — Adverse Event | 4 | 10 | 0
Not completed — Withdrawal by Subject | 9 | 8 | 0
Not completed — Lack of Efficacy | 6 | 7 | 0
Not completed — Lost to Follow-up | 0 | 4 | 0
Not completed — Protocol Violation | 0 | 4 | 0
Not completed — Pregnancy | 0 | 1 | 0
Period: Continuation Phase
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg | LTG XR, 250 mg | Baseline Failures
Started | 184 (83 and 101 participants from the 250 and 300 mg groups (DB Phase), respectively, entered the CP.) | 0 | 11 (See "Pre-assign. Details" for reasons why number starting CP does not equal number completing TP.)
Completed | 160 | 0 | 8
Not Completed | 24 | 0 | 3
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0
Not completed — Site Closed by Sponsor | 8 | 0 | 0
Not completed — Scheduling Error | 1 | 0 | 0
Not completed — Ran Out of Drug Due to Travel | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Phase: LTG XR, 300 mg: LTG XR, 300 mg/day in the Treatment phase
- Treatment Phase: LTG XR, 250 mg: LTG XR, 250 mg/day in the Treatment phase
- Total: Total of all reporting groups
Arm/Group | Treatment Phase: LTG XR, 300 mg | Treatment Phase: LTG XR, 250 mg | Total
Number analyzed (Participants) | 112 | 111 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (14.3) | 32.9 (12.6) | 33.4 (13.5)
Gender [Count of Participants; unit: Participants]
  Female | 56 | 66 | 122
  Male | 56 | 45 | 101
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 5 | 4 | 9
  Asian | 11 | 11 | 22
  Arabic/North African | 0 | 2 | 2
  White | 96 | 94 | 190
  Asian - Central/South Asian | 0 | 0 | 0
  Asian - East Asian | 0 | 0 | 0
Number of participants taking indicated concurrent antiepileptic drug at study entry [Number; unit: participants] — Antiepileptic drug (AED) being taken by participant at study entry; this characteristic is not applicable for the Continuation phase
  participants
    Valproate | 73 | 70 | 143
    Levetiracetam | 11 | 13 | 24
    Oxcarbazepine | 12 | 12 | 24
    Topiramate | 12 | 10 | 22
    Zonisamide | 3 | 5 | 8
    Pregabalin | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants in the 300 mg/Day Dose Group Who Prematurely Discontinued the Study Between Study Visit 5 (Approximately Week 7) and Visit 9 (End of the Treatment Phase)
Description: The percentage of participants prematurely discontinuing the study was calculated as the number of participants who discontinued the study divided by the number who reached Visit 5 minus major protocol violators. The Control group is composed of data from other similar studies and is not part of this study.
Time Frame: From Study Visit 5 through Visit 9 of the Treatment Phase (approximately Week 7 through Week 23)
Population: All randomized participants in the 300 mg/day dose group who began withdrawal of background antiepileptic drug (AED) (Visit 5) minus any major protocol violators
Measure: Number; unit: percentage of participants
Groups:
- Lamotrigine Extended-release (LTG XR), 300 mg: LTG XR, 300 mg/day
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg
Number analyzed (Participants) | 93
percentage of participants | 12

2. Secondary Outcome: The Percentage of Participants in the 250 mg/Day Dose Group Who Prematurely Discontinued the Study Between Study Visit 5 (Approximately Week 7) and Visit 9 (End of the Treatment Phase)
Description: The percentage of participants prematurely discontinuing the study was calculated as the number of participants who discontinued the study divided by the number who had reached Visit 5 minus major protocol violators. The Control group was composed of data from other similar studies and is not part of this study.
Time Frame: From Study Visit 5 through Visit 9 of the Treatment phase (approximately Week 7 through Week 23)
Population: All randomized participants in the 250 mg/day dose group who began withdrawal of background AED (Visit 5) minus any major protocol violators
Measure: Number; unit: percentage of participants
Arm/Group | LTG XR, 250 mg
Number analyzed (Participants) | 81
percentage of participants | 16

3. Secondary Outcome: Time to Discontinuation in the Treatment Phase
Description: Time (days) until the participant discontinued the study
Time Frame: From Study Visit 5 through Visit 9 of the Treatment phase (approximately Week 7 through Week 23)
Population: Intent-to-Treat (ITT) Population: All participants who were randomized and began dosing with study drug
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg | LTG XR, 250 mg
Number analyzed (Participants) | 112 | 111
Days | 147.3 (31.5) | 133.2 (45.6)

4. Secondary Outcome: Percentage of Participants Meeting Escape Criteria in the Treatment Phase
Description: The percentage of participants meeting Escape Criteria was calculated as the number of participants who met an Escape Criterion divided by the number who had reached Visit 5 minus major protocol violators. Escape Criteria are: (1) doubling of average monthly seizure frequency; (2) doubling of the highest consecutive 2-day seizure total; (3) occurrence of a new, more severe seizure type; or (4) worsening of generalized tonic-clonic seizures.
Time Frame: Study Visit 5 through Visit 9 of the Treatment phase (approximately Week 7 through Week 23)
Population: All randomized participants who began withdrawal of background AED (Visit 5) minus any major protocol violators
Measure: Number; unit: percentage of participants
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg | LTG XR, 250 mg
Number analyzed (Participants) | 93 | 81
percentage of participants | 4 | 6

5. Secondary Outcome: Percent Change From Baseline in Weekly Seizure Frequency Between Study Visits 3 (Start of Dosing) and 9 (End of the Treatment Phase)
Description: Change from Baseline was measured as the number of seizures at Visits 3 through 9 minus the number of seizures at Baseline. The number of partial seizures during treatment divided by the number of weeks of treatment was compared to the weekly seizure frequency during Baseline. A positive number equals a reduction in seizure frequency.
Time Frame: Baseline and Study Visit 3 through Visit 9 of the Treatment phase (Treatment Week 0 through Week 23)
Population: All randomized participants who began withdrawal of background AED (Visit 5) minus any major protocol violators
Measure: Median (Full Range); unit: percent change in seizures
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg | LTG XR, 250 mg
Number analyzed (Participants) | 93 | 81
percent change in seizures | 54.8 [-124.5 to 100.0] | 52.2 [-221.3 to 100.0]

6. Secondary Outcome: Number of Seizure-free Participants During the Last 12 Weeks of Treatment of the Treatment Phase
Description: The number of participants who had no seizures during the treatment period was calculated. The last 12 weeks of treatment were either Weeks 11-22 or 12-23 depending on which background AED was being withdrawn
Time Frame: The last 12 weeks of treatment of the Treatment phase (Monotherapy phase - approximately Week 11 through Week 23)
Population: All randomized participants who began withdrawal of background AED (Visit 5) minus any major protocol violators
Measure: Number; unit: participants
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg | LTG XR, 250 mg
Number analyzed (Participants) | 89 | 76
participants | 22 | 8

7. Secondary Outcome: Percent Change From Baseline in the Average Seizure Frequency Measured at the End of Participation in the Continuation Phase
Description: Change from baseline was calculated as the average seizure frequency at the end of the Continuation Phase minus the average seizure frequency at Baseline. The number of seizures during the Continuation phase divided by the number of weeks was compared to the number of seizures at Baseline. A positive number indicates a reduction in seizure frequency.
Time Frame: Baseline and start of Continuation phase through Week 24 or end of participation in the Continuation phase
Population: All participants who began the Continuation Phase
Measure: Median (Full Range); unit: percent change in seizures
Groups:
- Lamotrigine Extended-release (LTG XR), 300 mg: Treatment phase participants; LTG XR, 300 mg/day
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg | Baseline Failures
Number analyzed (Participants) | 184 | 11
percent change in seizures | 72.2 [-840.7 to 100.0] | 68.8 [-111 to 100]

8. Secondary Outcome: The Number of Participants With at Least the Specified Change in Seizure Frequency, Compared to Baseline, at the End of Participation in the Continuation Phase (Maximum of 24 Weeks)
Description: Change in seizure frequency was calculated as the average seizure frequency during the Continuation Phase minus the seizure frequency at Baseline.
Time Frame: Baseline and entire Continuation phase (24 Weeks)
Population: All participants who entered the Continuation Phase
Measure: Number; unit: participants
Arm/Group | Lamotrigine Extended-release (LTG XR), 300 mg | Baseline Failures
Number analyzed (Participants) | 184 | 11
participants
  At least a 25% reduction in seizures | 169 | 7
  At least a 50% reduction in seizures | 137 | 6
  At least a 75% reduction in seizures | 85 | 3
  100% reduction in seizures | 38 | 2
  At least a 50% increase in seizures | 6 | 3

ADVERSE EVENTS:
Description: For the Treatment phase, a frequency threshold of 5% in either treatment group was used. Because there are only 11 participants in the Baseline Failure group, only adverse events occurring in at least 3 participants in the 300 mg/day group are listed (1.6%).
Groups:
- Continuation Phase: LTG XR, 300 mg: Treatment phase participants; LTG XR, 300 mg/day
- Continuation Phase: Baseline Failures: Baseline failures that entered the Continuation Phase; LTG XR; 300 mg/day
Arm/Group | Treatment Phase: LTG XR, 300 mg | Treatment Phase: LTG XR, 250 mg | Continuation Phase: LTG XR, 300 mg | Continuation Phase: Baseline Failures
Serious Adverse Events (participants affected / at risk) | 3/112 | 5/111 | 3/184 | 1/11
Other Adverse Events (participants affected / at risk) | 44/112 | 52/111 | 47/184 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase: LTG XR, 300 mg (N=112) | Treatment Phase: LTG XR, 250 mg (N=111) | Continuation Phase: LTG XR, 300 mg (N=184) | Continuation Phase: Baseline Failures (N=11)
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Brain cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 1 | 0 | 0
Generalized seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Grand mal seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Periorbital hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 1
Upper GI bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase: LTG XR, 300 mg (N=112) | Treatment Phase: LTG XR, 250 mg (N=111) | Continuation Phase: LTG XR, 300 mg (N=184) | Continuation Phase: Baseline Failures (N=11)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 1
Dizziness (Nervous system disorders) | 12 | 10 | 11 | 2
Headache (Nervous system disorders) | 29 | 31 | 33 | 1
Insomnia (Psychiatric disorders) | 0 | 5 | 0 | 0
Nasalpharyngitis (Infections and infestations) | 7 | 7 | 5 | 0
Nausea (Gastrointestinal disorders) | 6 | 6 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 12 | 0 | 0
Somnolence (Nervous system disorders) | 5 | 6 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.